CLINICAL TRIAL: NCT01759017
Title: Molecular Imaging to Predict Response to Infliximab Therapy in Patients With Crohn's Disease
Brief Title: PET/CT to Predict Response to Infliximab Therapy in Patients With Crohn's Disease
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Paul Bernard Shyn, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2012P000570; BWH2012P000570 (Other: BWH)
Record Dates: First submitted 2012-12-21; First posted 2013-01-02 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Inflammatory bowel disease; IBD; Infliximab; PET; PET/CT
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infliximab responders: Gastroenterologist's overall assessment (response) Decrease in Harvey-Bradshaw index score of 2 or more points (clinical response) Harvey-Bradshaw index score less than 5 (clinical remission) Maintenance of steroid-free remission No Crohn's-related hospitalizations or surgeries
- Infliximab non-responders: Gastroenterologist's overall assessment (no response) Decrease in Harvey-Bradshaw index score of 1 or 0 points, or increase in HBI (no response) Harvey-Bradshaw index score greater than or equal to 5 (no remission) Resumption of steroid treatment Crohn's-related hospitalization or surgery

SUMMARY:
The costs and potential complications (side effects) of therapies currently used to treat Crohn's disease could be reduced if a non-invasive test existed that determined which therapies benefit patients and which do not. A non-invasive test is a test that does not involve cutting or entering the skin. Currently, once therapies are prescribed, doctors rely solely on clinical parameters to gauge whether the therapies are helpful. This includes evaluation of overall general well-being, abdominal pain, and number of liquid stools per day. There is no established and reliable non-invasive test that can predict whether a person is responding to therapy early in the course of treatment when these evaluations may be inconclusive.

During this research study we will look for changes in sugar metabolism on low-dose PET/CT before and 2 weeks after the first infusion of infliximab therapy. This is to find out if these changes can predict clinical response and steroid-free remission at two, six and 12 months, in patients with Crohn's disease.

DETAILED DESCRIPTION:
The costs and potential complications (side effects) of therapies currently used to treat Crohn's disease could potentially be reduced if a non-invasive test existed that determined which therapies benefit patients and which do not. Currently, once therapies are prescribed, doctors rely solely on clinical parameters to gauge whether the therapies are helpful. This includes evaluation of overall general well-being, abdominal pain, and number of liquid stools per day. There is no established and reliable non-invasive test that can predict whether a person is responding to therapy early in the course of treatment when these evaluations may be inconclusive.

During this research study we will look for changes in sugar metabolism on low-dose PET/CT before and 2 weeks after the first infusion of infliximab therapy. This is to find out if these changes can predict clinical response and steroid-free remission at two, six and 12 months, in patients with Crohn's disease.

PET/CT can be used to detect active inflammation (reaction of a part of the body to injury or infection) in Crohn's disease as well as complications such as ulcers, fissures, and strictures (thinning of, breaks in, and fixed narrowing of the bowel, respectively). PET (positron emission tomography) scans take pictures using special dyes that "light up" inside the body. This happens because the special dyes contain radiation, which is similar to the radiation in a standard x-ray. CT (computed tomography) uses x-rays and a computer to make pictures.

The radioactive tracer that will be used in this study is FDG. FDG is a radioactive sugar. FDG is approved by the U.S. Food and Drug Administration (FDA). This tracer can show early response to chemotherapy or other cancer treatments for a variety of tumors. Changes in FDG uptake accurately predict persistent response in as little as hours to days after therapy has begun. These changes often happen weeks to months before anatomic changes on CT or MRI. Sometimes the CT or MRI never changes.

One of the few FDG PET studies looking at treatment for an inflammatory condition showed that FDG uptake decreased significantly within two weeks of starting therapy for rheumatoid arthritis. Accurate early assessment with FDG PET/CT shortly after starting therapy with infliximab has the potential to change the standard clinical approach to both initial and continuing infliximab therapy in patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of symptomatic Crohn's disease or an established diagnosis of Crohn's disease with a suspected flare.
* Appropriate clinical candidate for infliximab induction therapy, as determined by the patient's gastroenterologist

Exclusion Criteria:

* Anti-TNF medications in the previous 6 months
* Pregnancy or plan to become pregnant
* Severe claustrophobia, sufficient to preclude PET/CT scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a new diagnosis of symptomatic Crohn's disease or an established diagnosis of Crohn's disease with suspected flare. The diagnosis of Crohn's disease will be based on the combination of clinical, imaging, endoscopic, and pathology findings.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Decrease in bowel FDG-uptake from enrollment to 2 weeks | one year
  Low-dose PET/CT will be performed at enrollment and at 2 weeks. Patients will be categorized as infliximab responders or non-responders based on clinical measures (overall assessment by the patient's gastroenterologist, Harvey-Bradshaw Index score, and any Crohn's-related hospitalization or surgery). We will determine if the decrease in bowel FDG-uptake is significantly different between responders and non-responders.

SECONDARY OUTCOMES:
Determination of the optimal threshold for decrease in FDG uptake on PET/CT for predicting clinical response | one year
  Using ROC analysis, we will determine the optimal threshold to separate patients classified as infliximab responders or non-responders for Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Shyn, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Shyn PB, Mortele KJ, Britz-Cunningham SH, Friedman S, Odze RD, Burakoff R, Goldberg JE, Erturk M, Silverman SG. Low-dose 18F-FDG PET/CT enterography: improving on CT enterography assessment of patients with Crohn disease. J Nucl Med. 2010 Dec;51(12):1841-8. doi: 10.2967/jnumed.110.080796. Epub 2010 Nov 15. PMID 21078803
- [Background] Shyn PB. 18F-FDG positron emission tomography: potential utility in the assessment of Crohn's disease. Abdom Imaging. 2012 Jun;37(3):377-86. doi: 10.1007/s00261-011-9793-y. PMID 21833729